CLINICAL TRIAL: NCT03366363
Title: Efficacy of Acupuncture Therapy Versus Sham Acupuncture on Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Acupuncture Therapy for Knee Osteoarthritis
Acronym: ATKOA Ⅱ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Collaborators: Beijing science and technology commission (Unknown)
Responsible Party: Principal Investigator, Ping Zhou, Clinical Professor, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017BL-077-01
Record Dates: First submitted 2017-11-20; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; acupuncture; electroacupuncture; sham acupuncture
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Acupuncturist (Electro-acupuncture group and Manual acupuncture group), Participant, Outcome Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electro-acupuncture (Experimental): 5 compulsory acupoints (ST35、EX-LE5、LR8、GB33 and Ashi) and 3 optional matching acupoints (stomach meridian syndrome：ST34、ST36、ST32、ST40、EX-LE2；gallbladder meridian syndrome：GB31、GB36、GB34、GB39、GB41；bladder meridian syndrome：BL39、BL40、BL57、BL60；San Yin meridian syndrome：LR7、SP9、SP10、KI10、SP4、SP6、LR3、KI3) will be chosen. Needles will be stimulated manually to achieve "De Qi" sensation and an electrical apparatus (Nanjing Jisheng Medical Co., Ltd., wave of 2/100Hz) will be then connected to the needles with alligator clips in pairs LR8-GB33 and two other matching acupoints. The stimulus intensity will be increased until the patient reports a strong but comfortable intensity. Patients will receive 30-minute, 24 sessions intervention over eight weeks.
  Interventions: Other: acupuncture
- manual acupuncture (Experimental): Participants in the manual acupuncture group have the same schedule as the Electro-acupuncture group except that the electrical apparatus has working power indicator and sound without actual current output.
  Interventions: Other: acupuncture
- sham acupuncture (Sham Comparator): Those in the sham acupuncture group receive shallow acupuncture at non-acupoints without manipulation，Deqi or actual current output.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — acupuncture is a therapy of traditional Chinese medicine，in which acupuncturist puncture the patient's skin at specific acupoints with needle.

SUMMARY:
Knee osteoarthritis (KOA), also called degenerative knee disease, is one of the most common bone and joint diseases in clinic. It was estimated to affect more than 9 million individuals in the United States in 2005 and is a leading cause of disability and medical costs. Most elderly people over the age of 65 have radiographic and/or clinical evidence of osteoarthritis. KOA is a lifelong disease which can lead to obvious pain, joint stiffness, limitation of activity and even joint failure or disability. Acupuncture is a popular treatment taken from ancient Chinese medicine, in which fine needles are placed into the body at specific points. Studies have shown that acupuncture can stimulate nerves under the skin, causing the body to produce natural pain-relieving substances (endorphins). However the evidences of acupuncture for KOA are contradictory. According to the review, intensive acupuncture with three sessions a week is more effective for KOA than sparse acupuncture with one session a week. Moreover, the papers published in the past years suggest that manual acupuncture and electro-acupuncture are most commonly used acupuncture therapy for the treatment of knee osteoarthritis. The aim of this study is to evaluate the efficacy of intensive electro-acupuncture or manual acupuncture versus sham acupuncture in reducing pain and improving function in patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75 years old, male or female
2. Single / bilateral knee pain, duration of more than 6 months
3. KL (Kellgren-Lawrence) grade Ⅱ or Ⅲ
4. NRS ≥ 4

Exclusion Criteria:

1. Surgery history of knee or waiting for surgery (knee replacement or knee arthroscopy)
2. Knee pain caused by other diseases (such as joint bodies, severe effusion of joint cavity, infection, malignant tumors, autoimmune diseases, trauma, fracture, gout, lumbosacral vertebrae disease, etc.)
3. History of arthroscopy within 1 year or intra-articular injection within 4 months
4. History of receiving acupuncture or massage treatment within 3 months
5. Severe acute/chronic organic or mental diseases
6. Coagulation disorders (such as hemophilia, etc.)
7. Cardiac pacemaker, metal allergy or needle phobia
8. Pregnant women, pregnant and lactating women
9. Participation in another clinical study in the past 3 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 8 weeks
  the percentage of patients with improvement in average pain (numerical rating scale, NRS) at least 2 units and in Western Ontario and Mcmaster Universities Osteoarthritis Index (WOMAC) function subscale score at least 6 units at 8 weeks. Pain NRS was a self-administered instrument, a number selected from 0-10 by participant. Intensity of pain range (over past week): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain. The WOMAC function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.

SECONDARY OUTCOMES:
Response rate | 16 weeks, 26 weeks
  the percentage of patients with improvement in average pain (numerical rating scale, NRS) at least 2 units and in Western Ontario and Mcmaster Universities Osteoarthritis Index (WOMAC) function subscale score at least 6 units at 16 and 26 weeks. Pain NRS was a self-administered instrument, a number selected from 0-10 by participant. Intensity of pain range (over past week): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain. The WOMAC function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.
Knee-joint pain | baseline, 8 weeks, 16 weeks and 26 weeks
  using numerical rating scale (NRS). NRS was a self-administered instrument, a number selected from 0-10 by participant. Intensity of pain range (over past week): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain.
Knee-joint pain | baseline, 8 weeks, 16 weeks and 26 weeks
  using WOMAC pain subscale. The WOMAC pain subscale referred to the patient's pain. It was comprised of 5 items, with each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst pain condition. An overall score range of 0 (minimum) to 20 (maximum), with higher scores indicating worse physical function.
Knee-joint function | baseline, 8 weeks, 16 weeks and 26 weeks
  using WOMAC function subscale. The WOMAC function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.
Knee-joint stiffness | baseline, 8 weeks, 16 weeks and 26 weeks
  using WOMAC stiffness subscale. The WOMAC stiffness subscale was comprised of 2 questions regarding the degree of stiffness experienced in the study knee. The WOMAC stiffness subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse stiffness. An overall score range of 0 (minimum) to 8 (maximum), with higher scores indicating more stiffness.
Quality of life | baseline, 8 weeks, 16 weeks and 26 weeks
  using 12-Item Short Form Health Survey. An overall score range of 0 (minimum) to 100(maximum), with higher scores indicating better quality of life.
Credibility score | 1 week（after the first treatment）
  using Credibility/expectancy questionnaire
Expectancy score | 1 week（after the first treatment）
  using Credibility/expectancy questionnaire
Blinding assessment | 4 weeks and 8 weeks
  Blinding assessment will be performed in all 9 centers
Global effect | 8 weeks, 16 weeks and 26 weeks
  Overall Treatment Effect (extremely improved, slightly improved, not changed, slightly aggravated, extremely aggravated)
Adverse events | first treatment up to 8 weeks
  Adverse Event Form

CONTACTS AND LOCATIONS:
Overall Officials: Cun-Zhi Liu, Study Chair — lcz623780@126.com
Locations (9):
- China (9):
  - Beijing Hostipal of Traditional Chinese Medicine affiliated to Capital medical University, Beijing, Beijing Municipality
  - Guang'an Men Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Beijing Hospital of Traditional Chinese and Western Medicine, Beijing, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Hospital of acupuncture-Moxibustion, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijin, Beijing Municipality
  - Affiliated Hospital of Hebei University of Chinese Medicine, Hebei, Hebei
  - First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tu JF, Yang JW, Shi GX, Yu ZS, Li JL, Lin LL, Du YZ, Yu XG, Hu H, Liu ZS, Jia CS, Wang LQ, Zhao JJ, Wang J, Wang T, Wang Y, Wang TQ, Zhang N, Zou X, Wang Y, Shao JK, Liu CZ. Efficacy of Intensive Acupuncture Versus Sham Acupuncture in Knee Osteoarthritis: A Randomized Controlled Trial. Arthritis Rheumatol. 2021 Mar;73(3):448-458. doi: 10.1002/art.41584. Epub 2021 Jan 15. PMID 33174383
- [Derived] Wang Q, Lv H, Sun ZT, Tu JF, Feng YW, Wang TQ, Liu CZ. Effect of Electroacupuncture versus Sham Electroacupuncture in Patients with Knee Osteoarthritis: A Pilot Randomized Controlled Trial. Evid Based Complement Alternat Med. 2020 Jul 30;2020:1686952. doi: 10.1155/2020/1686952. eCollection 2020. PMID 32802114
- [Derived] Tu JF, Yang JW, Wang LQ, Wang Y, Li JL, Zhang N, Lin LL, Yu ZS, Liu CZ. Efficacy of electro-acupuncture and manual acupuncture versus sham acupuncture for knee osteoarthritis: statistical analysis plan for a randomized controlled trial. Trials. 2019 Jul 4;20(1):394. doi: 10.1186/s13063-019-3513-2. PMID 31272488
- [Derived] Tu JF, Yang JW, Lin LL, Wang TQ, Du YZ, Liu ZS, Hu H, Zhao JJ, Yu XG, Jia CS, Wang J, Wang T, Hou YQ, Zou X, Wang Y, Shao JK, Wang LQ, Yu ZS, Liu CZ. Correction to: Efficacy of electro-acupuncture and manual acupuncture versus sham acupuncture for knee osteoarthritis: study protocol for a randomised controlled trial. Trials. 2019 Apr 10;20(1):204. doi: 10.1186/s13063-019-3338-z. PMID 30971318
- [Derived] Tu JF, Yang JW, Lin LL, Wang TQ, Du YZ, Liu ZS, Hu H, Zhao JJ, Yu XG, Jia CS, Wang J, Wang T, Hou YQ, Zou X, Wang Y, Shao JK, Wang LQ, Yu ZS, Liu CZ. Efficacy of electro-acupuncture and manual acupuncture versus sham acupuncture for knee osteoarthritis: study protocol for a randomised controlled trial. Trials. 2019 Jan 25;20(1):79. doi: 10.1186/s13063-018-3138-x. PMID 30683147